CLINICAL TRIAL: NCT04867239
Title: Temporal Changes of Metabolic Indicators and Quality of Life by a Two-day Patient Education Program for Metabolic Syndrome Patients
Brief Title: A Two-day Education Program for Metabolic Syndrome Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sang Yeoup Lee, Professor, Pusan National University Yangsan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 05-2014-039
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic Syndrome; Motivation; Patient Education; Quality of Life
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A two-day education program (Other): During the camp, the multidisciplinary team provided disease information, lifestyle modification, nutrition, and exercise for metabolic syndrome. Participants visited at 3- and 6-month after camp for follow-up.
  Interventions: Other: A two-day education progra

INTERVENTIONS:
Other: A two-day education progra — During the camp, the multidisciplinary team provided disease information, lifestyle modification, nutrition, and exercise.

SUMMARY:
This study was to evaluate the temporal change of metabolic indicators and quality of life by a two-day patient education program.

DETAILED DESCRIPTION:
This study aimed to evaluate whether a two-day multidisciplinary education camp comprising doctors, nurses, exercise instructors, dietitians, social workers, and health administrators could initiate healthy lifestyle habits, improve health markers though lifestyle modification, increase knowledge and understanding of the disease, and have a profitable effect on mental health in relation to depression and quality of life for patients with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* people satisfied with metabolic syndrome criteria

Exclusion Criteria:

* None

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-05-23 (Actual); Primary Completion 2014-11-23 (Actual); Study Completion 2014-11-30 (Actual)

PRIMARY OUTCOMES:
Waist circumference (cm) | Change from pre-camp at 3-month and 6-month after camp
  Change in waist circumference at 3-month and 6-month after camp
Blood pressure (mmHg) | Change from pre-camp at 3-month and 6-month after camp
  Change in blood pressure at 3-month and 6-month after camp
Korean version of EuroQol-5D (the minimum-maximum value, 0-1) | Change from pre-camp at 3-month and 6-month after camp
  Change in score of Korean version of EuroQol-5D at 3-month and 6-month after camp. Higher scores mean a better outcome.
Korean version of Beck depression inventory-II (the minimum-maximum value, 0-63) | Change from pre-camp at 3-month and 6-month after camp
  Change in score of Korean version of Beck depression inventory-II at 3-month and 6-month after camp. Higher scores mean a worse outcome.
Korean version of Beck anxiety inventory (the minimum-maximum value, 0-63) | Change from pre-camp at 3-month and 6-month after camp
  Change in score of Korean version of Beck anxiety inventory at 3-month and 6-month after camp. Higher scores mean a worse outcome.
Nutritional knowledge score (the minimum-maximum value, 0-20) | Change from pre-camp at 3-month and 6-month after camp
  Change in nutritional knowledge score at 3-month and 6-month after camp. Higher scores mean a better outcome.
Total cholesterol (mg/dL) | Change from pre-camp at 3-month and 6-month after camp
  Change in total cholesterol (mg/dL) level at 3-month and 6-month after camp
Triglyceride (mg/dL) | Change from pre-camp at 3-month and 6-month after camp
  Change in triglyceride (mg/dL) level at 3-month and 6-month after camp
HDL cholesterol (mg/dL) | Change from pre-camp at 3-month and 6-month after camp
  Change in HDL cholesterol (mg/dL) level at 3-month and 6-month after camp
LDL cholesterol (mg/dL) | Change from pre-camp at 3-month and 6-month after camp
  Change in LDL cholesterol (mg/dL) level at 3-month and 6-month after camp

CONTACTS AND LOCATIONS:
Overall Officials: Sang Yeoup Lee, MD, PhD, Principal Investigator — Pusan National University Yangsan Hospital